CLINICAL TRIAL: NCT06793852
Title: Investigation of the Effect of Shoulder Pain on Joint Position Sense, Postural Control, Tactical Sensory and Muscle Strength in Chronic Hemiplegic Patients
Brief Title: Shoulder Pain and Its Effects on Joint Position, Strength, Tactical Sensory and Posture in Hemiplegia
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, PT, PhD, Karabuk University
Other Study IDs: shoulder pain in stroke
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-01

CONDITIONS: Hemiplegic Shoulder Pain
Keywords: Stroke; Pain; Postural Control; Sensation; Muscle Strength
MeSH Terms: conditions — Stroke; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- participants with shoulder pain
- participants without shoulder pain

SUMMARY:
The main purpose of this study is to reveal the effects of shoulder pain in chronic hemiplegic patients with a more comprehensive and holistic perspective through evaluation and correlation methods. It is thought that these evaluations can make significant contributions to the understanding of the etiology and treatment of post-stroke shoulder pain. The focus of the study is to deeply examine the effects of shoulder pain on joint position sense, postural control, tactile sense and muscle strength in chronic hemiplegic patients.

DETAILED DESCRIPTION:
This study aims to investigate the effects of shoulder pain on joint position sense, postural control, tactile sensation, and muscle strength in chronic hemiplegic stroke patients. Designed as a cross-sectional descriptive study, it involved participants divided into two groups based on the presence or absence of shoulder pain. The assessments included joint position sense , postural control , tactile sensation , gross grip strength, and pinch grip strength . The findings of this study are expected to contribute to clinical practice by aiding in the development of more effective interventions for managing post-stroke shoulder pain. Additionally, it aims to serve as a foundation for future comprehensive research, emphasizing the critical role of addressing pain in the rehabilitation process.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months post-stroke, diagnosis of hemiplegia after stroke, aged 18 or older, having cognitive abilities and cooperation required to fulfill the study requirements, and willingness to participate in the study.

Exclusion Criteria:

* cognitive impairment interfering with informed consent or adherence to study assessments, aphasia, the presence of major neurological or rheumatological diseases affecting the musculoskeletal system other than stroke, and a history of surgery on the affected shoulder prior to stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals diagnosed with stroke and receiving treatment at the Special Safranbolu Special Education and Rehabilitation Center in Karabük province. Based on previous similar studies, the sample size was calculated using power analysis with 80% power and a significance level of α=0.05, resulting in 78 participants.
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
inclinometer | Baseline
Postural Assessment Scale for Stroke Patients (PASS-T) | Baseline
Semmes-Weinstein Monofilament test | Baseline
dynamometer | Baseline
pinchmeter | Baseline

SECONDARY OUTCOMES:
Personal information form | Baseline
Visual Analog Scale | Baseline
Shoulder Pain and Disability Index | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson RD, Chae J. Hemiplegic Shoulder Pain. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):641-55. doi: 10.1016/j.pmr.2015.06.007. Epub 2015 Sep 9. PMID 26522903